CLINICAL TRIAL: NCT04133623
Title: Ibuprofen Versus Ketorolac by Mouth in the Treatment of Acute Pain From Osteoarticular Trauma: a Randomized Double-blind Controlled Study.
Brief Title: Ibuprofen Versus Ketorolac by Mouth in the Treatment of Acute Pain From Osteoarticular Trauma
Acronym: IbuKet
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RC 21/18
Record Dates: First submitted 2019-10-18; First posted 2019-10-21 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2022-01

CONDITIONS: Acute Pain Due to Trauma
Keywords: osteoarticular acute pain; ketorolac; ibuprofen
MeSH Terms: interventions — Ketorolac; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: double dummy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketorolac (Experimental): Administration of ketorolac 0.5 mg/kg up to 10 mg, one single dose at the enrollment. This group will receive also a placebo indistinguishable from the ibuprofen.
  Interventions: Drug: Ketorolac
- Ibuprofen (Active Comparator): Administration of ibuprofen 10 mg/kg up to 600 mg, one single dose at the enrollment. This group will receive also a placebo indistinguishable from the ketorolac.
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Ketorolac — Administration of ketorolac 0.5 mg/kg up to 10 mg, one single dose at the enrollment. This group will receive also a placebo indistinguishable from the ibuprofen.
  Arms: Ketorolac
Drug: Ibuprofen — Administration of ibuprofen 10 mg/kg up to 600 mg, one single dose at the enrollment. This group will receive also a placebo indistinguishable from the ketorolac.
  Arms: Ibuprofen

SUMMARY:
Pain is the leading cause of access to the paediatric emergency department (ED) and present in up to 78% of cases.

Acute osteoarticular traumatic pain is often treated inadequately, and there is little data about the best treatment for children. The ibuprofen and ketorolac are respectively the most used and one of the most powerful NSAIDs. In literature, there is no direct comparison between those two medications.

The objective of the study depends on the level of pain:

* in severe traumatic acute pain (>=7 points): to evaluate if ketorolac is superior to ibuprofen in the treatment of pain (n=130 children, 65 allocated to ketorolac and 65 to ibuprofen)
* in moderate traumatic acute pain (<7 points): to evaluate if ibuprofen is not inferior to ketorolac in the treatment of pain (n=120 children, 60 allocated to ketorolac and 60 to ibuprofen)

ELIGIBILITY:
Inclusion Criteria:

* Age between 8 and 18 years
* Moderate to severe pain (value>= 4 on the Numerical Rating scale / NRS)
* Pain due to a trauma at limbs that has occurred in the last 48 hours

Exclusion Criteria:

* Administration of any analgesic in the previous 8 hours.
* Allergy known to one of the active ingredients
* Known hepatopathy or nephropathy
* Suspicion of violence by others
* Chronic use of painkillers
* Inability to report pain due to the presence of: intellectual disability (IQ <70); moderate-severe hearing loss; communication limitations such as patient mutism; unable to write; inability to speak Italian
* Chronic neurological or metabolic diseases,
* Positive history for ease of bleeding, coagulation disorder or
* thrombocytopenia
* A history of gastritis or esophagitis in the last 30 days
* Multiple trauma
* Vascular-vascular deficit
* State of pregnancy

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 212 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Pain reduction assessed on the NRS scale 60 minutes after the administration of the drug | 60 minutes after the administration of the drug
  NRS scale will be asked after 60 minutes from the administration of the drug. To evaluate the NRS scale the patient is asked to express how much pain he feels through a number ranging from 0 to 10 in which 10 is the maximum pain. This is one of the most used methods in pain assessment.
  The difference will be calculated from the baseline.

SECONDARY OUTCOMES:
NRS 30 minutes after the administration of the drug | 30 minutes after the administration of the drug
  NRS scale will be asked after 30 minutes from the administration of the drug. To evaluate the NRS scale the patient is asked to express how much pain he feels through a number ranging from 0 to 10 in which 10 is the maximum pain. This is one of the most used methods in pain assessment.
NRS at time 90 minutes after the administration of the drug | 90 minutes after the administration of the drug
  NRS scale will be asked after 90 minutes from the administration of the drug. To evaluate the NRS scale the patient is asked to express how much pain he feels through a number ranging from 0 to 10 in which 10 is the maximum pain. This is one of the most used methods in pain assessment.
NRS at time 120 minutes after the administration of the drug | 120 minutes after the administration of the drug
  NRS scale will be asked after 120 minutes from the administration of the drug. To evaluate the NRS scale the patient is asked to express how much pain he feels through a number ranging from 0 to 10 in which 10 is the maximum pain. This is one of the most used methods in pain assessment.
Patients who obtain a value of NRS <4 after 30 minutes from the administration of the drug. | 30 minutes after the administration of the drug
  NRS scale will be asked after 30 minutes from the administration of the drug. To evaluate the NRS scale the patient is asked to express how much pain he feels through a number ranging from 0 to 10 in which 10 is the maximum pain. This is one of the most used methods in pain assessment.
Patients who obtain a value of NRS <4 after 60 minutes from the administration of the drug | 60 minutes after the administration of the drug.
  NRS scale will be asked after 60 minutes from the administration of the drug. To evaluate the NRS scale the patient is asked to express how much pain he feels through a number ranging from 0 to 10 in which 10 is the maximum pain. This is one of the most used methods in pain assessment.
Patients who obtain a value of NRS <4 after 90 minutes from the administration of the drug. | 90 minutes after the administration of the drug
  NRS scale will be asked after 90 minutes from the administration of the drug. To evaluate the NRS scale the patient is asked to express how much pain he feels through a number ranging from 0 to 10 in which 10 is the maximum pain. This is one of the most used methods in pain assessment.
Patients who obtain a value of NRS <4 after 120 minutes from the administration of the drug. | 120 minutes after the administration of the drug.
  NRS scale will be asked after 120 minutes from the administration of the drug. To evaluate the NRS scale the patient is asked to express how much pain he feels through a number ranging from 0 to 10 in which 10 is the maximum pain. This is one of the most used methods in pain assessment.
Patients who obtain a reduction of NRS of more than 3 points after 30 minutes from the administration of the drug. | NRS scale will be asked after 30 minutes from the administration of the drug.
  30 minutes after the administration of the drug.
Patients who obtain a reduction of NRS of more than 3 points after 60 minutes from the administration of the drug. | 60 minutes after the administration of the drug.
  NRS scale will be asked after 60 minutes from the administration of the drug. To evaluate the NRS scale the patient is asked to express how much pain he feels through a number ranging from 0 to 10 in which 10 is the maximum pain. This is one of the most used methods in pain assessment
Patients who obtain a reduction of NRS of more than 3 points after 90 minutes from the administration of the drug. | 90 minutes after the administration of the drug.
  NRS scale will be asked after 90 minutes from the administration of the drug. To evaluate the NRS scale the patient is asked to express how much pain he feels through a number ranging from 0 to 10 in which 10 is the maximum pain. This is one of the most used methods in pain assessment.
Patients who obtain a reduction of NRS of more than 3 points after 120 minutes from the administration of the drug | 120 minutes after the administration of the drug.
  NRS scale will be asked after 120 minutes from the administration of the drug. To evaluate the NRS scale the patient is asked to express how much pain he feels through a number ranging from 0 to 10 in which 10 is the maximum pain. This is one of the most used methods in pain assessment
Adverse effects in the two groups | within 120 minutes from the administration of the drug
  By the medical or nursing staff patients will be evaluated after administration of the drug (headache, nausea, vomiting, somnolence, dyspepsia, abdominal pain, pruritus, dizziness and other reported symptoms).
Emergency department outcome | within 120 minutes from the administration of the drug
  Number of children that, following the emergency department visit, are:
  1. discharged at home
  2. temporary observed in the emergency department
  3. hospitalized

CONTACTS AND LOCATIONS:
Overall Officials: Barbi Egidio, MD PhD, Study Chair — Institute for Maternal and Child Health IRCCS Burlo Garofol
Locations (3):
- Italy (3):
  - Azienda Ospedaliera Santa Maria degli Angeli, Pordenone
  - Institute for Maternal and Child Health - IRCCS Burlo Garofolo-, Trieste
  - Ospedale Santa Maria della Misericordia, Udine

REFERENCES:
- [Derived] Ghirardo S, Trevisan M, Ronfani L, Zanon D, Maestro A, Barbieri F, De Nardi L, Amaddeo A, Barbi E, Cozzi G. Oral ibuprofen versus oral ketorolac for children with moderate and severe acute traumatic pain: a randomized comparative study. Eur J Pediatr. 2023 Feb;182(2):929-935. doi: 10.1007/s00431-022-04759-3. Epub 2022 Dec 17. PMID 36526794